CLINICAL TRIAL: NCT07364292
Title: Shared Decision Making in Dialysis Modality Selection: a Lived Experience From Nephrologists. A Nationwide Qualitative Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Anne-Lorraine Clause, Medical doctor in nephrology, Erasme University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SRB2023343
Record Dates: First submitted 2024-01-28; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: End Stage Renal Disease
Keywords: shared-decision-making; dialysis modality selection; kidney failure; home-based therapies
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: explanatory study using mixed method qualitative data analysed systematically by quantitative method (Q method)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nephrologists (Other): no other arm
  Interventions: Behavioral: Q methodology

INTERVENTIONS:
Behavioral: Q methodology — Q- sorting operation is done during a face-to-face meeting of the participant and the interviewer. Participants rank-order a set of statements or opinions into a grid. They rank the importance of statements relative to all others. A specific characteristic of Q Sort is that participants are forced to prioritize amongst statements. During the ranking procedure, they must explain their reasoning process on their positioning of their cards ("thinking-aloud" their reasoning). This audiotaping of the thinking aloud during the actual completion of the Q-Sort allows to not only gain insights in the perceptions of the participants, but also in their underlying reasoning, emotions, and motivation.

SUMMARY:
International guidelines for kidney failure emphasize the importance of aligning renal replacement therapy (RRT) modality selection with individuals' preferences through high-quality, structured education. However, observational qualitative studies suggest that pre-dialysis education remains inconsistently delivered, with substantial centre-to-centre variation in the content and organization of Belgian pre-dialysis programs despite a shared healthcare policy.

Multiple barriers to home-based therapies have been repeatedly reported at both the unit and patient levels, including nursing shortages, limited availability of trained staff, financial constraints, high rates of unplanned dialysis initiation, distress at treatment start, low health literacy, and an increasingly frail and comorbid patient population.

Yet, a minority of dialysis units appear able to mitigate these barriers more effectively than others. This discrepancy raises concern that centre-oriented priorities (unit throughput, cost-effectiveness, technical performance) may still outweigh patient-centred goals (supporting life priorities and meaningful shared decision-making).

This study aims to explore nephrologists' beliefs, knowledge, and attitudes regarding shared decision-making in dialysis modality selection and their potential influence on the adoption of alternative RRT modalities beyond in-centre hemodialysis. Q methodology will be used to capture and compare shared viewpoints and patterns of disagreement across participants.

DETAILED DESCRIPTION:
Objective: To explore the nephrologist's lived experience regarding shared-decision making during dialysis decision making process.

Design: Prospective, monocentric, interventional, mixed-methods design (qualitative and quantitative) using Q methodology.

Rationale:

International guidelines related to kidney failure strongly support individuals' preferences when choosing their renal replacement modality through appropriate education provision. However, previous observational qualitative studies have shown that pre-dialysis education is poorly delivered, with wide centre-to-centre variation in the content and organization of Belgian pre-dialysis programs, despite a shared healthcare policy.

Many logistical issues raised as "barriers" at the centre level, but also at the patient level, have already been identified in previous studies: shortage of nurses, lack of trained staff in home-based treatment or education provision, limited financial resources, a high rate of unplanned patients, patient distress at dialysis initiation, a high rate of poor health literacy, and a shift in patient mix toward higher rates of comorbidities and frailty are the most frequently cited barriers.

However, some (a minority of) dialysis units succeed in solving part of these common issues, while most do not, suggesting that nephrologists and healthcare providers may not have all the clues or the vision of care to overcome these factors. This raises concerns about the primacy of a centre-oriented culture (unit management, cost-effectiveness, technical achievements) rather than prioritizing a patient-centred approach (meeting patients' therapeutic and life goals and actively engaging them in the modality decision-making process).

Within this explanatory research project, the primary objective is to explore in-depth insights into the perspective (beliefs and attitude) of healthcare professionals regarding dialysis decision making process.

The expected first benefit is a better understanding of individual behaviours, values, beliefs, and expectations regarding the implementation of shared decision-making in dialysis modality selection, as well as areas of consensus and disagreement surrounding this controversial topic.

Indeed, a lack of structured educational programs and national guidelines to support healthcare professionals in educating end-stage kidney disease patients is observed in many European countries and likely contributes to the low adoption rates and variable penetration of home-based treatments, as well as pre-emptive transplantation and conservative care.

Methods and analysis:

Investigators are using Q-sort methodology as the foundation for semi-structured interviews. Q-sort combines qualitative and quantitative approaches to measure subjectivity, such as opinions and beliefs. Unlike interviews, it assesses consensus and disagreement among individuals on a specific topic. The process involves creating a set of statements (Q-set) that capture the diversity of scientific or public opinions on that particular topic. Participants (P-set) then rank these statements based on their agreement using a forced-choice grid. Correlations are analyzed between participants' Q-sorts to identify shared perspectives within the group. This study is reported according to the Consolidated criteria for reporting qualitative research (COREQ) guidelines (12).

Study population:

Investigators are using maximum variation sampling. Twenty-five active nephrologists were purposively selected to represent diverse ages, dialysis and home dialysis experience, and gender perspectives nationwide. Dialysis units were chosen to represent different program sizes and organizational cultures. All participants gave written informed consent.

Data collection:

Investigators are using a Q-sort methodology involving the forced ranking of predefined actions in response to each clinical case vignette (Supplemental material). In total, four clinical vignettes, each with nine potential actions, were created based on the literature and consensus within the research team. In a pilot phase, all statements were assessed for clarity and absence of ambiguity. During the sorting process, a think-aloud approach was employed to elicit participants' reasoning behind their classifications, followed by a 30-minute semi-structured interview guided by the Q-sorts.

All sessions were conducted by two authors, audiotaped, and transcribed verbatim.

Q methodology is used to systematically study subjectivity-that is, subjective opinions, values, or beliefs-to answer questions about "how" and "what." It allows the identification of shared viewpoints on a topic, revealing areas of consensus and disagreement.

Correlations between participants, rather than correlations between measures, are explored; thus, the analysis correlates Q-sorts and provides indications of similar segments of subjectivity within the participant group. A post-sort interview, or "think-aloud" reasoning, is provided by respondents during or immediately after the Q-sort to explain their reasoning during the ranking process.

A structured approach, based on prior hypotheses or a literature review suggesting that the quality and content of pre-dialysis programs are influenced by several key factors, will be used. Thematic analysis includes:

1. interest, expectations, and involvement of nephrologists and nurses in pre-dialysis care;
2. emphasis on meaningful activities and life goals rather than modality-related technical aspects;
3. level of perceived patient-related prejudice hindering true shared decision-making;
4. transparency regarding all available options;
5. service provision around alternative modalities.

Demographic data such as age, gender, academic work, peritoneal dialysis or home hemodialysis experience (in years), as well as overall professional experience of each participant, will be collected, analyzed, and reported.

ELIGIBILITY:
Inclusion Criteria:

* nephrologists professionnaly active

Exclusion Criteria:

* non active or retired nephrologists
* nephrologist who do not have regular contact with ESKD patients or who do not engage in treatment discussion

Ages: 30 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Number of distinct Q-methodology viewpoints (factors) identified from nephrologists' Q-sorts related to shared decision-making in dialysis modality choice, as derived from Q-factor analysis. | Time Frame: Once, at the baseline study visit (single Q-sort session), up to 90' per participant
  Q-sort data will be collected using a forced-ranking of predefined actions in response to clinical vignettes. The primary quantitative endpoint is the number of interpretable factors extracted from participants' Q-sorts using principal component factor analysis with varimax rotation.
  Results will be reported as:
  * Number of factors identified (count),
  * Number (%) of participants significantly loading on each factor (p < 0.01)
  * Factor loadings (correlation coefficients) per factor reported as mean (SD) and range.

SECONDARY OUTCOMES:
Number and content of overarching themes and sub-themes identified from semi-structured interviews relevant to dialysis-decision making. | Once, during the baseline session (up to 30 minutes per participant)
  Semi-structured interviews (think-aloud and post-sort interview) will be audio-recorded, transcribed verbatim, and analyzed using thematic analysis with a phenomenological approach.
  Outcomes will be reported as:
  * Number of overarching themes identified (count),
  * Number of sub-themes within each overarching theme (count),
  * Thematic domains related to shared decision-making (SDM) in dialysis modality selection.

CONTACTS AND LOCATIONS:
Locations (1):
- HUB Erasme, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Allen K, Shaw KL, Spry JL, Dikomitis L, Coyle D, Damery S, Fotheringham J, Lambie M, Williams IP, Davies S. How does organisational culture facilitate uptake of home dialysis? An ethnographic study of kidney centres in England. BMJ Open. 2024 Dec 27;14(12):e085754. doi: 10.1136/bmjopen-2024-085754. PMID 39732481
- [Background] Brown EA, Brivio GB, Van Biesen W. Towards a better uptake of home dialysis in Europe: understanding the present and looking to the future. Clin Kidney J. 2024 Jun 5;17(Suppl 1):i3-i12. doi: 10.1093/ckj/sfae082. eCollection 2024 May. PMID 38846418
- [Result] Cortvrindt C, Van Biesen W, Gambino G, Clause AL. Factors influencing renal replacement therapy modality choice from the nephrologist's perspective. J Nephrol. 2024 Apr;37(3):635-645. doi: 10.1007/s40620-024-01915-w. Epub 2024 Mar 21. PMID 38512379